CLINICAL TRIAL: NCT01709656
Title: A Molecule Basic Study of Early Warning for New Pathogenic Risk of Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gu Jieruo, Department of Rheumatology, Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: [2012]2-31
Record Dates: First submitted 2012-10-10; First posted 2012-10-18 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSC plus NSAID (Experimental): human mesenchymal stem cells:1*10^4-6 cells /Kg , IV (in the vein) on day 1 of each 14-60 day cycle,1-6 times treatment, plus non-steroid anti-inflammatory drugs (NSAID: "celecoxib", "Celebrex®" 0.2g Bid(twice a day),PO (Per Os).
  Duration of treatment:24 weeks for follow up. collect peripheral blood (PBMCs and serums)of those patients at baseline and every 4 weeks for basic study after they signed informed consent.
  Interventions: Biological: MSC; Drug: "celecoxib", "Celebrex®"
- NSAID (Experimental): non-steroid anti-inflammatory drugs (NSAID: "celecoxib", "Celebrex®" 0.2g Bid(twice a day),PO (Per Os);a total of 24 weeks for follow up;collect peripheral blood (PBMCs and serums)of those patients at baseline and every 4 weeks for basic study after they signed informed consent.
  Interventions: Drug: "celecoxib", "Celebrex®"

INTERVENTIONS:
Biological: MSC — human mesenchymal stem cells,1*10^4-6 cells /Kg , IV (in the vein) on day 1 of each 14-60 day cycle,1-6 times treatment.
  a total of 24 weeks for follow up.
  Arms: MSC plus NSAID
Drug: "celecoxib", "Celebrex®" — non-steroid anti-inflammatory drugs (NSAID):"celecoxib", "Celebrex®" 0.2g Bid(twice a day),PO (Per Os);a total of 24 weeks for follow up

SUMMARY:
The investigators will recruit active ankylosing spondylitis patients for injection treatment of Human Mesenchymal Stem Cells (a prospective, open-label, masculine medicine controlled(NSAIDs), clinical trial), and collect their Peripheral Blood Lymphocyte (PBMCs) and sera before and after the treatment of 24 weeks to test the gene expression profiles and study related pathogenesis of AS

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 16-65 years, sign the Informed Consent
2. Fulfill 1984 modified NewYork classification criteria for AS
3. Have an active refractory disease defined by a score ≥40 on the Bath AS Disease Activity Index (BASDAI) (0-100) despite optimal non-steroidal anti-inflammatory drug (NSAID) treatment.
4. Commitment to contraceptive for woman

Exclusion Criteria:

1. Completely stiff spine
2. Received spinal or joint surgery within 2 months
3. Received anti-TNF therapy within 3 months
4. History of the listed diseases: heart failure, Multiple sclerosis, severe chronic obstructive pulmonary disease, frequent infections, lymphoma or other cancers, tuberculosis
5. Female of pregnancy or breast feeding
6. Hb≤ 9g/dl for male or Hb ≤ 8.5 g/dl for male, ALT/AST≥2folds of upper level normal range, Creatine≥120mol/L(≤1.4mg/dl)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the proportion of patients which disease activity reaches ASAS(assessment in ankylosing Spondylitis)20 remission criteria | 24 weeks

SECONDARY OUTCOMES:
BASDAI score comparing to baseline | 24 weeks
BASFI score comparing to baseline | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, M.D., Principal Investigator — Department of Rheumatology , Third Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Department of Rheumatology, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China